CLINICAL TRIAL: NCT04674397
Title: Effect of Donor Nephrectomy on Markers of Bone Function in Living Kidney Donors
Brief Title: BOne Dysfunction in Donor NEphrectomieS
Acronym: BONES
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: R03728
Record Dates: First submitted 2020-03-16; First posted 2020-12-19 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Renal Failure; Kidney Donors
Keywords: Donor; CKD-MBD; FGF23
MeSH Terms: conditions — Renal Insufficiency; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Urine and DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group: Living kidney donors
  Interventions: Radiation: Radioisotope GFR test

INTERVENTIONS:
Radiation: Radioisotope GFR test

SUMMARY:
Most dialysis patients die from vascular disease, which is statistically associated with changes related to chronic kidney disease associated mineral bone disorder (CKD-MBD)3-9. Understanding the mechanisms behind this high death rate is crucial to improving the length and quality of life for patients with all grades of kidney disease, including those on dialysis. This is a priority for patients and clinicians alike.

Most humans with early CKD are asymptomatic and unaware that they have a problem with their kidneys. Therefore they are unlikely to consult a doctor and early CKD is often unrecognised. Patients who are aware of early CKD often have other co-morbidities including diabetes, hypertension and vascular disease which, in the setting of a clinical study, complicate the identification of changes solely resulting from CKD. However over the past decade living kidney donation has become increasingly common and is now the source of organs for more than 120 patients annually at Manchester's renal transplant centre. Prospective donors are carefully examined and known to have normal kidney function without other co-morbidities. They then undergo a planned unilateral nephrectomy and lose approximately 50% of their kidney mass, creating an immediate state of moderate CKD. Over subsequent months the remaining kidney will hypertrophy and partially correct this, although the mechanisms are unknown. In the immediate post-operative period donors are inpatients on the kidney transplant ward and have regular blood and urine tests meaning that careful study of metabolic processes during their recovery is relatively easy by analysis of serial plasma and urine samples. Sequential changes in the plasma and urine levels of different bone turnover markers and metabolites can be analysed and will provide valuable new information to increase our understanding of the initial stage of CKD-MBD development.

DETAILED DESCRIPTION:
The likelihood of five year survival for a 60 year old dialysis patient (50%) is significantly worse than for breast (88%), prostate (90%) or colon cancer sufferers (56%)1, but robust information about the contributory risk-factors to inform clinician-patient discussions is lacking2. Most dialysis patients die from vascular disease, which is statistically associated with changes related to chronic kidney disease associated mineral bone disorder (CKD-MBD)3-9. Understanding the mechanisms behind this high death rate is crucial to improving the length and quality of life for patients with all grades of kidney disease, including those on dialysis. This is a priority for patients and clinicians alike.

A recent Kidney Disease Improving Global Outcomes (KDIGO) statement highlighted the poor level of understanding of the mechanisms of CKD-MBD in early and late kidney disease which inhibits the development of targeted therapies to either halt the process or at least improve outcomes10-12.

CKD confers certain atypical risk factors for mortality, most notably a state of disordered mineral metabolism which is implicated in the development of hyperphosphataemia, hyperparathyroidism and vascular calcification. Despite the variety of biological malfunctions attributed to CKD-MBD, the pathophysiology is not understood, partly because there is no animal model of progressive CKD. Rodent models do not survive long enough for the all changes of CKD-MBD to develop. Therefore current therapy is inadequate, and usually deployed late in the course of CKD when the patient has progressed to end-stage renal disease. Furthermore there is no reliable evidence that current therapies improve patient outcome in terms of length or quality of life. The progression of CKD is not always linear and less than 5% of patients proceed to end-stage renal disease. While aetiology of renal impairment determines progression to some extent, there is no reliable means of determining who will progress and who will not so that targeted study of early CKD-MBD pathogenesis is not possible.

Most humans with early CKD are asymptomatic and unaware that they have a problem with their kidneys. Therefore they are unlikely to consult a doctor and early CKD is often unrecognised. Patients who are aware of early CKD often have other co-morbidities including diabetes, hypertension and vascular disease which, in the setting of a clinical study, complicate the identification of changes solely resulting from CKD. However over the past decade living kidney donation has become increasingly common and is now the source of organs for more than 120 patients annually at Manchester's renal transplant centre. Prospective donors are carefully examined and known to have normal kidney function without other co-morbidities. They then undergo a planned unilateral nephrectomy and lose approximately 50% of their kidney mass, creating an immediate state of moderate CKD. Over subsequent months the remaining kidney will hypertrophy and partially correct this, although the mechanisms are unknown. In the immediate post-operative period donors are inpatients on the kidney transplant ward and have regular blood and urine tests meaning that careful study of metabolic processes during their recovery is relatively easy by analysis of serial plasma and urine samples. Sequential changes in the plasma and urine levels of different bone turnover markers and metabolites can be analysed and will provide valuable new information to increase our understanding of the initial stage of CKD-MBD development.

ELIGIBILITY:
Inclusion Criteria:

Potential living kidney donors who have completed the medical assessment and have been accepted for kidney donation. -

Exclusion Criteria:

1. Known to have a significant pathology that may influence markers of renal/bone axis - including but not limited to thyroid disorders, parathyroid disorders, amputees, Paget's disease, and severe osteoporosis.
2. Previous treatment with bisphosphonates or denosumab.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: living kidney donors
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in renal volume post-donation | 1 month
  Volume of the remaining kidney is measured by serial MRI scans pre-donation, 4-7 days post-donation and 1 month post donation
Change in kidney function post-donation | 3 months
  isotope GFR is measured 1 month after donation; serum creatinine estimated GFR is measured at pre-donation, 30 minutes, 60 minutes, Day 1,2,3,4 and 7, 2 weeks, 3 weeks, 1 month, 2 months and 3 months after donation; Serum cystatin C estimated GFR is measured at pre-donation, Day 7 and 1 month after donation.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No